CLINICAL TRIAL: NCT02188667
Title: An Integrative and Sustainable Approach to Pain Management in Primary Care
Brief Title: Integrating Patient Reported Outcomes (I-PRO) Study for Multidisciplinary Pain Care
Acronym: I-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201300433; 8578749 (Other Grant/Funding Number: Pfizer, Inc.)
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Noncancer Pain
Keywords: Chronic Noncancer Pain; Musculoskeletal Pain; Neuropathic Pain; Headache Pain
MeSH Terms: conditions — Musculoskeletal Pain; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Providers of Novel Care (Active Comparator): Providers in the treatment group will be asked (1) to complete a series of six online education modules in pain care, (2) will be given access to new patient reported outcomes questionnaire data collected from patients within the electronic health record, (3) asked to review this data and related care recommendations during the patient visit, and (4) asked to complete baseline and monthly online surveys related to experiences and satisfaction with providing care to patients with chronic noncancer pain.
  Interventions: Other: Providers of Novel Care
- Providers of Usual Care (Sham Comparator): Providers in the control group will provide care as usual to patients and will be asked to complete baseline and monthly online surveys related to experiences and satisfaction with providing care to patients with chronic noncancer pain.
  Interventions: Other: Providers of Usual Care

INTERVENTIONS:
Other: Providers of Novel Care — Providers in the treatment group will be asked (1) to complete a series of six online education modules in pain care, (2) will be given access to new patient reported outcomes questionnaire data collected from patients within the electronic health record, (3) asked to review this data and related care recommendations during the patient visit, and (4) asked to complete baseline and monthly online surveys related to experiences and satisfaction with providing care to patients with chronic noncancer pain.
  Arms: Providers of Novel Care
Other: Providers of Usual Care — Providers in the control group will provide care as usual to patients and will be asked to complete baseline and monthly online surveys related to experiences and satisfaction with providing care to patients with chronic noncancer pain.
  Arms: Providers of Usual Care

SUMMARY:
The purpose of this study is to assess the impact of clinician education, electronic health record integrated patient reported outcomes, and electronic health record integrated decision support on pain-related care quality, outcomes, and service utilization.

DETAILED DESCRIPTION:
The initiative has three components to aid clinicians' care of patients with chronic noncancer pain: (1) education, (2) standardized patient reported outcomes data collection, and (3) evidence-based brief treatment reminders. Practices will be randomized to either receive the three novel components (treatment group) or continue with usual care (control group).

Providers in the treatment group will be asked (a) to complete a series of six online education modules in pain care, (b) will be given access to new patient reported outcomes questionnaire data collected from patients within the electronic health record, (c) asked to review this data and related care recommendations during the patient visit, and (d) asked to complete baseline and monthly online surveys related to experiences and satisfaction with providing care to patients with chronic noncancer pain.

Providers in the control group will provide care as usual to patients and will be asked to complete baseline and monthly online surveys related to experiences and satisfaction with providing care to patients with chronic noncancer pain.

Primary study outcomes include comparison of treatment and control group provider and patient satisfaction surveys. Secondary outcome measures include provider referral rates, patient outcomes, patient treatments recommended/ordered, and patient service utilization/costs.

ELIGIBILITY:
Inclusion Criteria:

* Providers at one of six active Community Health and Family Medicine locations in the University of Florida Health system Gainesville service area (Hampton Oaks, Eastside, Jonesville, and Haile) between May 1, 2014 and September 1, 2015
* Doctor of Medicine (MD), Doctor of Osteopathic Medicine (DO), Advanced Registered Nurse Practitioner (ARNP), Physician Assistant (PA) or other faculty professional providing primary care services

Exclusion Criteria:

* Residents or other trainees at one of four active Community Health and Family Medicine locations in the University of Florida Health system Gainesville service area (Hampton Oaks, Eastside, Jonesville, and Haile) between May 1, 2014 and September 1, 2015

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Provider Satisfaction Survey | Up to 15 months
  This is a 16 item web based questionnaire about general experiences and satisfaction with providing care to patients with chronic noncancer pain. Data will be collected at baseline (June 2014) and monthly thereafter through the end of the study period (July 2014 - September 2015). Provider satisfaction data for both the treatment and control groups will be compared.
Patient Satisfaction Survey | Up to 15 months
  This is a four to five question phone survey (depending on whether patient is seeing a provider in a treatment or control group) about general and pain-specific satisfaction with visit. Data will be collected after each visit for chronic noncancer pain through the study period (July 2014 - September 2015). Patient satisfaction data for both the treatment and control groups will be compared.

SECONDARY OUTCOMES:
Hospital Readmission Rates | Up to 5 years
  The data will be collected retrospectively for a history of hospital readmission rates (June 2011 - June 2014). Once the new care model starts for the clinicians, data will be collected at baseline (July 2014) and at the end of the study period (September 2015) for an indication of trends. Data for both the treatment and control groups will be compared.
Lab Orders and Results | Up to 5 years
  The data will be collected retrospectively for a history of lab orders and results (June 2011 - June 2014). Once the new care model starts for the clinicians, data will be collected at baseline (July 2014) and at the end of the study period (September 2015) for an indication of trends. Data will be
Prescribed and Dispensed Medications | Up to 5 years
  The data will be collected retrospectively for a history of prescribed and dispensed medications (June 2011 - June 2015). Once the new care model starts for the clinicians, data will be collected at baseline (July 2014) and at the end of the study period (September 2015) for an indication of trends. Data for both the treatment and control groups will be compared.
Pain Intensity | Up to 5 years
  The data will be collected retrospectively for a history of pain intensity (June 2011 - June 2014). Once the new care model starts for the clinicians, data will be collected at baseline (July 2014) and at the end of the study period (September 2015) for an indication of trends. Data for both the treatment and control groups will be compared.
Medical Costs | Up to 5 years
  The data will be collected retrospectively for a history of medical costs (June 2011 - June 2014). Once the new care model starts for the clinicians, data will be collected at baseline (July 2014) and at the end of the study period (September 2015) for an indication of trends.This will include cost of pain related care for charge amounts and billed amounts for specialist services, hospital services, and utilization of non-physician services (e.g., pharmacy, physical therapy, etc.). Data for both the treatment and control groups will be compared.
Health Care Utilization | Up to 5 years
  The data will be collected retrospectively for a history of health care utilization (June 2011 - June 2014). Once the new care model starts for the clinicians, data will be collected at baseline (July 2014) and at the end of the study period (September 2015) for an indication of trends. This will include utilization of specialist services, hospital services, and utilization of non-physician services (e.g., pharmacy, physical therapy, etc.). Data for both the treatment and control groups will be compared.
Pain Specialist Referral Rates | Up to 5 years
  The data will be collected retrospectively for a history of pain specialist referral rates (June 2011 - June 2014). Once the new care model starts for the clinicians, data will be collected at baseline (July 2014) and at the end of the study period (September 2015) for an indication of trends. Data for both the treatment and control groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Harle, PhD, Principal Investigator — University of Florida; Robert W Hurley, MD, PhD, Principal Investigator — University of Florida; Nicole Marlow, PhD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - Family Medicine at Hampton Oaks, Gainesville, Florida
  - Family Medicine at Haile Plantation, Gainesville, Florida
  - Eastside Community Practice, Gainesville, Florida
  - Family Medicine at Jonesville, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided